CLINICAL TRIAL: NCT02644785
Title: Investigation of Anaphylactic Reaction in Cases Undergoing Cardiac By-Pass Surgery
Brief Title: Serum Tryptase Levels During Cardiac Surgery, Diagnosis and Treatment Decisions for Allergic Reactions
Status: Completed | Type: Observational
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, MENEKSE OKSAR, Assistant Professor, Mustafa Kemal University
Other Study IDs: 2014/10
Record Dates: First submitted 2015-12-24; First posted 2016-01-01 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2016-02

CONDITIONS: Protamine Allergy; Protamine Adverse Reaction
Keywords: cardiac by-pass; protamine; tryptase; hypotension; anaphylaxis
MeSH Terms: conditions — Hypotension; Anaphylaxis | interventions — Protamines; glucosulfone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: protamine — Protamine infusion exposures
  Other Names: promin

SUMMARY:
The investigators aim to assess tryptase test efficacy for measuring the allergic response to protamine during cardiac bypass surgery. Additionally, the investigators aim to establish a differential diagnosis on the basis of potential allergens or clinical causes.

DETAILED DESCRIPTION:
Venous blood samples from cardiac surgery cases will be obtained for tryptase measurement upon admission to the operating room (OR) and immediately prior to and 30 min after protamine infusion initiation. A rapid effect-response-based clinical assessment will be made using clinical and laboratory monitoring data for diagnosis and treatment decisions during protamine infusion, which may complicate the recovery from surgery.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac by-pass cases

Exclusion Criteria:

* Insulin dependent diabetes
* Atopy
* Drug allergy history

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elective cardiac By-Pass surgery cases
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Patients number with high tryptase level (> 25 µg/L ). | 30 min
  Tryptase will be measured using the ImmunoCAP Tryptase kit (Phadia, Uppsala, Sweden), and the cutoff level for elevated tryptase is >11.5 µg/L. A 25 µg/L cutoff value has been found to be highly suggestive of an İmmunoglobulin E (IgE) -mediated reaction.

SECONDARY OUTCOMES:
Patients number with allergic reaction involving of 1 or more organ/systems (skin, respiratory, or cardiovascular system) following the study drug infusion. In this study, mainly the cardiovascular and skin symptoms will be focused on. | 30 min
  These outcomes will be determined following the Council for International Organizations of Medical Sciences (CIOMS 1999 and ) definitions for anaphylactic reactions. Additionally, (World Health Organization - Uppsala Monitoring Centre) WHO-UMC system will be used for assesment of causality categories for adverse drug reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Menekse Oksar, M.D., Principal Investigator — Mustafa Kemal University Medical School
Locations (1):
- Mustafa Kemal University Hospital, Antakya, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Krishna MT, York M, Chin T, Gnanakumaran G, Heslegrave J, Derbridge C, Huissoon A, Diwakar L, Eren E, Crossman RJ, Khan N, Williams AP. Multi-centre retrospective analysis of anaphylaxis during general anaesthesia in the United Kingdom: aetiology and diagnostic performance of acute serum tryptase. Clin Exp Immunol. 2014 Nov;178(2):399-404. doi: 10.1111/cei.12424. PMID 25070464
- [Result] Malinovsky JM, Decagny S, Wessel F, Guilloux L, Mertes PM. Systematic follow-up increases incidence of anaphylaxis during adverse reactions in anesthetized patients. Acta Anaesthesiol Scand. 2008 Feb;52(2):175-81. doi: 10.1111/j.1399-6576.2007.01489.x. Epub 2007 Nov 13. PMID 18005384
- [Result] Mertes PM, Laxenaire MC, Alla F; Groupe d'Etudes des Reactions Anaphylactoides Peranesthesiques. Anaphylactic and anaphylactoid reactions occurring during anesthesia in France in 1999-2000. Anesthesiology. 2003 Sep;99(3):536-45. doi: 10.1097/00000542-200309000-00007. PMID 12960536
- See also: The authors reported that elevated acute serum tryptase (>141% from baseline or absolute tryptase >15.7 mg/L) is highly predictive of IgE-mediated anaphylaxis and that these two methods of interpretation are comparable. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Krishna+MT%2C+York+M%2C+Chin+T%2C+et+al%3A+Multi-centre+retrospective+analysis+of+anaphylaxis+during+general+anaesthesia+in+the+United+Kingdom%3A+aetiology+and+diagnostic+performance+of+acute+serum+tryptase.+Clin+Exp+Immunol+178%3A399-404%2C+2014
- See also: Malinovsky et al. reported that tryptase concentrations were elevated in 50% of their patients, and the positive and negative predictive values (PPV and NPV) of tryptase were 100% for both tryptase >12 and >25 at the first samples. — http://www.ncbi.nlm.nih.gov/pubmed?term=malinovskyjm,decagnys,wesself,etal.systematicfollow-upincreasesincidenceofanaphylaxisduringadversereactionsinanesthetizedpatientsactaanaesthesiascand52175-181,2008&cmd=correctspelling
- See also: Krishna et al. reported sensitivities, specificities, PPV and NPV for a tryptase of >25 mcg/L to be 64, 74, 82 and 52 respectively in 103 patients which were similar to the values reported by Mertes et al. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Mertes+Anesthesiology+2003%3B99%3A536-45